CLINICAL TRIAL: NCT07138976
Title: Comparison of Safety and Effectiveness Between Endoscopic Ultrasound-guided and Ultrasound-guided Pancreatic Biopsy in Focal Pancreatic Disease: A Multi-center, Retrospective, Propensity Score Analysis
Brief Title: EUS- and US- Guided Biopsy for Pancreatic Lesion
Status: Not yet recruiting | Type: Observational
Sponsor: Tian'an Jiang (Other)
Responsible Party: Sponsor-Investigator, Tian'an Jiang, Tian'an Jiang, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Other Study IDs: Pancreatic biopsy-PSM
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sampling tissue — EUS- and US- guided pancreatic biopsy

SUMMARY:
Endoscopic ultrasound (EUS) and ultrasound (US) are the two primary imaging modalities used to guide pancreatic needle biopsy. This study aimed to compare the diagnostic performance and complications associated with EUS- and US-guided pancreatic biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Between January 2017 and December 2023, 2663 consecutive patients with focal pancreatic disease underwent 2729 procedures for pancreatic tissue acquisition from focal pancreatic lesions at seven university teaching hospitals in China.

Exclusion Criteria:

* Patients were excluded from the study if they had less than 12 months of follow-up, were lost to follow-up, had incomplete follow-up data, or underwent intraoperative biopsy or fluid aspiration.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with focal pancreatic disease underwent procedures for pancreatic tissue acquisition
Sampling Method: Non-Probability Sample
Enrollment: 2517 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic inaccuracy | 1-year

DOCUMENTS (1):
  • Study Protocol (2025-08-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT07138976/Prot_000.pdf